CLINICAL TRIAL: NCT05879653
Title: A Phase 2, Open-label, Multi-institutional Study to Evaluate the Efficacy of Induction Therapy With MK-3475 and ASG-22CE Followed by Radiation Therapy With MK-3475 in Patients With MIBC Who Are Unfit for or Refuse Radical Cystectomy
Brief Title: Pembrolizumab and EV With Radiation Therapy for MIBC Patients (PEVRAD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyoto University Hospital (Other)
Collaborators: University of Tsukuba (Other); Osaka Metropolitan University (Other); Kobe City Medical Center General Hospital (Unknown); Merck Sharp & Dohme LLC (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Takashi Kobayashi, Professor, Kyoto University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IACT21079
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer
Keywords: Bladder preservation; Radiation therapy; Immunotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; enfortumab vedotin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MK-3475 and ASG-22CE With Radiation Therapy (Experimental)
  Interventions: Drug: MK-3475; Drug: ASG-22CE; Procedure: maximal TURBT; Radiation: Radiation therapy

INTERVENTIONS:
Drug: MK-3475 — During the induction phase, MK-3475 200 mg will be administered as four cycles of 3-weeks regimen, with ASG-22CE 1.25 mg/kg administered on Day 1 and Day 8 of each cycle. The treatment and maintenance phases will consist of 9 cycles of one course per 6 weeks, with MK-3475 400 mg administered on Day 1 of each course at Q6W.
  Other Names: Pembrolizumab
Drug: ASG-22CE — During the induction phase, four cycles of 3-weeks regimen are administered, with ASG-22CE 1.25 mg/kg administered on Day 1 and Day 8 of each cycle.
  Other Names: Enfortumab vedotin
Procedure: maximal TURBT — All participants who were not determined to have PD on imaging during the induction phase should have had a maximal TURBT performed at 13 (± 1week) weeks after the first dose of trial drug.
Radiation: Radiation therapy — Radiotherapy will be initiated no later than 8 weeks after maximal TUR-BT. In this trial, a total dose of 56 Gy will be delivered using 2 Gy per dose. 40 Gy/20 fr (2 Gy/fr) to the small pelvis followed by 16 Gy /8 fr (2 Gy/fr) to the whole bladder 5 times a week for 5 consecutive days using Three-Dimensional Conformal Radiation Therapy (3D-CRT).

SUMMARY:
This study is designed to assess the efficacy and safety of induction therapy with MK-3475 and ASG-22CE and radiation therapy with MK-3475 in patients with cT2-4aN0M0 muscle invasive bladder cancer who are unfit for or refuse radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Male/female participants who are at least 18 years of age on the day of signing informed consent and who have a first confirmed diagnosis of MIBC with predominant urothelial histology obtained via a diagnostic or maximal TURBT within 90 days prior to enrollment.

     Note: Participants with mixed histology are eligible provided the urothelial component is ≥50%.
  2. Has clinically non-metastatic bladder cancer (N0M0) determined by imaging (CT of the chest and CTU/MRU of abdomen and pelvis), assessed by the site.
  3. Male participants:

     A male participant must agree to use a contraception and not to donate sperm during the administration of MK-3475 and ASG-22CE and for at least 90 days after the last dose of MK-3475 and for 6 months after ASG-22CE.
  4. Female participants:

     A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
     1. Not a woman of childbearing potential (WOCBP) OR
     2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of MK3475 and for 6 months after ASG-22CE and RT.
  5. The participant provides written informed consent for the trial.
  6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
  7. Demonstrates adequate organ function. All screening laboratory tests should be performed within 10 days prior to the first dose of study intervention.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Has the presence of diffuse CIS (multiple foci [4 or greater] of CIS) throughout the bladder.
2. Has the presence of UC at any site outside of the urinary bladder in the previous 2 years except for Ta/T1/CIS of the upper tract if the patient has undergone a complete nephroureterectomy.
3. Has the presence of any small cell or neuroendocrine component in the tumor tissue sample.
4. Has a known additional malignancy that is progressing or has required active therapy within the past 3 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or other carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) who have undergone potentially curative therapy are not excluded. Participants with low-risk prostate cancer (T1-T2a, Gleason score ≤6, and PSA <10 ng/mL) either treated with definitive intent any time before screening or untreated in active surveillance are not excluded.
5. Has limited bladder function with frequency of small amounts of urine (< 30 mL), urinary incontinence, or requires self-catheterization or a permanent indwelling catheter.
6. Has a history of radiation therapy to the pelvic region for any reason.

   Prior/Concomitant Therapy
7. Has received prior pelvic/local radiation therapy or any antineoplastic treatment for MIBC.

   Note: Prior treatment for NMIBC with intravesical instillation therapy such as BCG or intravesical chemotherapy is permitted, but must be completed ≥28 days before the first dose of the trial drug. Prior systemic treatment received for treatment of NMIBC is not permitted.
8. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
9. Has received prior therapy with an ASG-22CE or other MMAE-containing ADCs.
10. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

    Note: please refer to Section 5.5 for information on COVID-19 vaccines Prior/Concurrent Clinical Study Experience
11. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 3 months before the first dose of study intervention.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

    Diagnostic Assessments
12. A WOCBP who has a positive urine pregnancy test within 72 hours prior to the first dose of study intervention (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Has uncontrolled diabetes. Uncontrol diabetes is defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7% to <8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
14. Has ongoing sensory or motor neuropathy Grade 2 or higher.
15. Has active keratitis or corneal ulceration. Subjects with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator.
16. Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease, with a 1-week washout, is permitted.
17. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial drug.
18. Has severe hypersensitivity (≥Grade 3) to MK-3475, ASG-22CE and/or any of their excipients.
19. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid).
20. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
21. Has an active infection requiring systemic therapy.
22. Has a known history of Human Immunodeficiency Virus (HIV) infection. The test should be performed within 28 days prior to the first dose of the trial drug.
23. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. The test should be performed within 28 days prior to the first dose of the trial drug.
24. Has not adequately recovered from major surgery or has ongoing surgical complications.
25. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
26. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
27. Pregnant or lactating, or female patients or male patients who wish to become pregnant from the time of screening to 120 days after the last dose of MK-3475 and 6 months after radiotherapy and the last dose of ASG-22CE, or their partners.
28. Has had an allogenic tissue/solid organ transplant.
29. Has a documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with NYHA Class IV within 6 months prior to the first dose of the trial drug.
30. Or, if participation in this clinical trial is considered inappropriate according to the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Bladder Intact Event-Free Survival (BI-EFS) rate | 2 years
  To evaluate bladder intact event-free survival (BI-EFS) rate at 2 year after study enrollment assessed by cystoscopy, cytology, biopsy results by central pathology review, and imaging evaluation.

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) Rate at 38 weeks | 38 weeks
  The pathologic complete response rate is based on the central pathology review of tumor bed biopsies performed at 38 weeks and the results of imaging studies performed by each institution.
Overall Survival (OS) | 2 years
  OS is defined as the time from study enrollment to death from any cause.
Metastasis-Free Survival (MFS) | 2 years
  Metastasis-free survival is defined as the time from study enrollment to the first documented evidence of nodal or distant metastases as assessed by CT of chest and CTU or MRU of the abdomen and pelvis and/or biopsy results assessed by central pathology review, or death from any cause. If biopsy is not feasible due to participant safety, the imaging alone will be sufficient.
Number of participants who experienced an adverse event (AE) | 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be presented.
Number of participants who discontinued study intervention due to an AE | 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.
Change from Baseline in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline and up to approximately 2years
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. The change from baseline in Global Health Status/Quality of Life (EORTC QLQ-C30 Items 29 and 30) combined score will be presented.
Change from Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | Baseline and up to approximately 2years
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a better quality of life. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score will be presented.
Change from Baseline in Urinary, Bowel, and Sexual Domains of the Bladder Cancer Index (BCI) | Baseline and up to approximately 2years
  The BCI is a validated, condition-specific health questionnaire assessing quality of life among participants with bladder cancer. The BCI contains 36 items which assess 3 domains (urinary, bowel, and sexual) with function and bother subdomains. Scores range from 0 to 100 with higher scores corresponding to better functioning and health-related quality of life. The change from baseline in the combined scores of the urinary, bowel, and sexual domains of the BCI will be presented.
Change from Baseline in the Visual Analog Score (VAS) of the European Quality of Life (EuroQoL)-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) | Baseline and up to approximately 2years
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 cm vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". The change from baseline in EQ-5D-5L VAS will be presented.
Time to Deterioration (TTD) in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the EORTC QLQ-C30 | 2 years
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. TTD in Global Health Status/Quality of Life is defined as the time from baseline to the first onset of a 10 point or greater decrease from baseline in the Global Health Status/Quality of Life (EORTC QLQ-C30 Items 29 and 30) combined score, with or without subsequent confirmation.
TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | 2 years
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a better quality of life. TTD in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score is defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in physical functioning Items 1 to 5 scale scores.
TTD in Urinary, Bowel, and Sexual Domains of the BCI | 2 years
  The BCI is a validated, condition-specific health questionnaire assessing quality of life among participants with bladder cancer. The BCI contains 36 items which assess 3 domains (urinary, bowel, and sexual) with function and bother subdomains. Scores range from 0 to 100 with higher scores corresponding to better functioning and health-related quality of life. TTD in BCI is defined as a 6, 7, and 7 points or greater worsening from baseline for urinary, bowel, and sexual domains, respectively, with or without subsequent confirmation, under a right-censoring rule.
TTD in the VAS of the EQ-5D-5L | 2 years
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 cm vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". TTD in EQ-5D-5L VAS is defined as the time from baseline to the first onset of a 7 point or greater decrease from baseline in EQ-5D-5L VAS, with or without subsequent confirmation, under a right-censoring rule.

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kobayashi, MD,PhD, Principal Investigator — Kyoto University Hospital
Locations (4):
- Japan (4):
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kyoto University Hospital, Kyoto, Kyoto
  - Osaka Metropolitan University Hospital, Osaka, Osaka

IPD SHARING:
Plan to Share IPD: No